CLINICAL TRIAL: NCT03893864
Title: Bioavailability and Impact of the Administration of Coenzyme Q10, on Mitochondrial Function Associated With Exercise Under Stress Conditions in Physically Active Individuals of Senescence Age
Brief Title: Bioavailability and Impact of Coenzyme Q10 in Stressing Exercise in Senescence Athletes
Acronym: CoQ10Sport
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre d'Alt Rendiment (Other)
Collaborators: Hospital Sant Joan de Deu (Other); University of Barcelona (Other); Indena S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CAR-2018 CoQ10
Record Dates: First submitted 2019-03-05; First posted 2019-03-28 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Coenzyme Q10; Oxidative Stress; Aging
Keywords: Coenzyme Q10; Ubiquinone; Ubiquinol; Oxidative pattern; Exercise
MeSH Terms: conditions — Motor Activity | interventions — coenzyme Q10

STUDY DESIGN:
Intervention Model Description: Interventional study of 22 subjects, 12 under supplemental intervention and 10 as control subjects. Both groups are similar subjects with same characteristics and condition. The interventional group will receive a supplementaction of CoQ10 (100 mg) during one month, the Control group nothing.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The participants of the interventional group know they are taking a nutritional supplementation in study to improve health condition. Only the outcome evaluators, blood analisis, exercise testing data processing, muscle biopy analisys do not know if the samples come from control or interventional group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (CoQ10) (Experimental): Runner athletes > 50 years old, took 100 mg/d of fitosomed Ubiquinone with lunch, daily, during one month, maintaining their usual training sessions
  Interventions: Dietary Supplement: Administration of a product with Fitosomed Ubiquinone; Procedure: Coenzyme Q10 level in muscle biopsies; Diagnostic Test: Coenzyme Q10 level in plasma, blood cells, urine cells; Diagnostic Test: Total antioxidant capacity after strenous exercise
- Control Group (Active Comparator): Runner athletes > 50 years old with the same characteristics as the Experimental arm, served as control group, maintaining the training sessions Both groups were evaluated before and after the month of intervention or no intervention.
  Interventions: Diagnostic Test: Coenzyme Q10 level in plasma, blood cells, urine cells; Diagnostic Test: Total antioxidant capacity after strenous exercise

INTERVENTIONS:
Dietary Supplement: Administration of a product with Fitosomed Ubiquinone — Healthy runner athletes, > 50 years old, without any chronic illness, without any other nutritional supplementation or drug intervention, took 100 mg/d of fitosomed Ubiquinone with lunch, daily, during one month, maintaining their usual training sessions.
  Other Names: Coenzyme Q10; UbiQuisome
  Arms: Intervention Group (CoQ10)
Procedure: Coenzyme Q10 level in muscle biopsies — Determination of the muscle Ubiquinone concentration, the metabolic and structure characteristics of the muscle before and after one month of supplementation
  Other Names: Muscle Biopsy
  Arms: Intervention Group (CoQ10)
Diagnostic Test: Coenzyme Q10 level in plasma, blood cells, urine cells — Determination of Ubiquinone concentration in different tissues before and after one month of supplementation or not
Diagnostic Test: Total antioxidant capacity after strenous exercise — Determination of the Total Antioxidant Capacity after strenous exercise in the Climate Chamber
  Other Names: TAC after exercise

SUMMARY:
It is proposed to establish a group of subjects composed of 10 healthy individuals of> 50 years and <65, physically active, without metabolic or inflammatory pathology. All of them will undergo a health examination and the physical condition and the absence of contraindication of the sports practice will be characterized through a monitored effort test. Each subject will take a capsule of coenzyme Q10® INDENA for 30 days. The dose to be administered is 100 mg/d of CoQ10 a with food (noon). The state of physical condition and the biochemical and biological variables that reflect oxidative stress and mitochondrial functioning before and after the intervention will be measured.

DETAILED DESCRIPTION:
The purpose of the study is in the first time determine the variation of the levels of coenzyme Q10 in different tissues, plasma, urinary epithelium, muscle, mononuclear cells, before and after the administration during one month of 100 mg of phytosomal ubiquinone (INDENA). Secondly, it is intended to determine the antioxidant functionality of the administered ubiquinone, evaluating its effect on the oxidative pattern that occurs after an exercise of moderate intensity, but performed in a stressful environment, a climatic chamber where the temperature is 35ºC and there is 55% humidity. To this end, the collaboration of 12 healthy volunteers, and 10 control subjects, over 50 and under 65, active runners with experience, without active inflammatory pathology, without prescribed medical treatment and with the commitment not to take any nutritional supplementation. There is also a compromise by athletes on maintaining the diet and training as it is at the time of the first evaluation The subjects sign an informed consent to carry out the study and they are shown the acceptance of the Ethics Committee approved by the General Directorate of Sports of the Generalitat of Catalonia. Basal blood samples are taken, the sample is taken from the first urine in the morning and a muscle biopsy is performed on the vastus lateralis of the m. quadricipitalis. On a second day, a progressive, maximum effort test is carried out in order to characterize the level of physical condition and determine the working regimes in the climatic chamber. They are re-scheduled for a third day for that purpose. On that day blood is drawn to obtain the Total Antioxidant Capacity of the blood and they are exposed to the temperature and humidity and are asked to run on the treadmill for 5 minutes at each of the speeds corresponding to 70, 75 and 80% of the maximum speed reached in the first test. At the end a lactate sample is taken. This period of 15 minutes is repeated 3 times. When finished, at the 30th minute, a new blood sample is taken to assess the TAC postexercise/exposition.

The stress test and blood extractions, urine collection and muscle biopsy are repeated after one month of taking the phytosomed Ubiquinone.

There is a control group of 10 subjects who follow absolutely the same path, but do not take any supplementation (Ubiquinone) and do not have a muscle biopsy.

ELIGIBILITY:
Inclusion criteria

* Athletes over 50 active at this time
* Runners
* Without medical treatment
* Without acute or chronic inflmatory disease
* No recent infectious processes
* No muscle or joint injuries in the last 6 months
* Stable training during the evaluation period
* Without taking supplementation

Exclusion criteria

* Injuried, sickness, during the study
* Lack of compromise
* Inflamatory process
* Abandon the training by any reason

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Change in the concentration of CoQ10 on different tissues after supplementation for a month | 6 months
  Evaluate the change in the concentration of CoQ10 on plasma, muscle, monouclear cells and urinary epithelium, by specific analysis of every sample tissue at the Pathology Dept and the Methabolopathies Dept of the Pediatric Hospital of Sant Joan de Deu

SECONDARY OUTCOMES:
Effect of the CoQ10 supplementation on the oxidative response to stressing exercise under heat and humidity | 3 months
  Determination of the inflammatory response before and after stressing exercise at the climate chamber at 35ºC and 55% humidity. The procedure is by the analysis of the venous blood extracted previous the exercise stress and 30 minutes after the period of work
Effect of the CoQ10 supplementation on the inflammatory response to stressing exercise under heat and humidity | 3 months
  Determination of the Total antioxidant capacity before and after stressing exercise at the climate chamber at 35ºC and 55% humidity. The procedure is by the analysis of the venous blood extracted previous the exercise stress and 30 minutes after the period of work

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Artuch, MD, PhD, Study Chair — Hospital Sant Joan de Deu, Barcelona
Locations (1):
- Centre D'Alt Rendiment, Sant Cugat, Sant Cugat Del Vallés, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No